CLINICAL TRIAL: NCT06164158
Title: Role of Procedural Videos in Teaching the Surgery Residents: A Randomized Control Trial
Brief Title: Role of Procedural Videos in Teaching the Surgery Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Mansoor Ahmed, Principal Investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ShaheedZABMU123
Record Dates: First submitted 2023-11-21; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Educational Techniques; Surgical Procedure, Unspecified

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Half were made to watch the procedural videos and learn the steps of the procedure and then made to perform procedure
  Interventions: Other: Procedural Videos
- Control Group (Experimental): Other half group did not watch the procedural videos and were made to perform procedure.
  Interventions: Other: No procedural videos

INTERVENTIONS:
Other: Procedural Videos — A randomized controlled trial was conducted at Pakistan Institute of Medical Sciences (PIMS) Islamabad between September 1, 2023 to November 30, 2023 under ethical approval from the Institutional ethical review board.
  Arms: Study Group
Other: No procedural videos — No procedural videos
  Arms: Control Group

SUMMARY:
A randomized controlled trial was conducted at Pakistan Institute of Medical Sciences (PIMS) Islamabad after approval from the Institutional ethics review board. Fifty-four surgical residents in training and who have completed at least 3 months of surgical training were enrolled in the study. After the residents had performed the procedure initially, 27 were made to watch the procedural videos and learn the steps of the procedure while those of the other group did not watch the videos. Participants of both the groups were made to perform the procedure. GARS (global assessment rating score) was calculated for each individual during their second procedure. All procedures were performed under the supervision of a consultant surgeon who was blinded about the groups and make assessment of the GARS (global assessment rating score).

DETAILED DESCRIPTION:
This study was conducted in 2 phases. In Phase-I just after the enrollment, all the residents performed the procedure from which initial GARS (global assessment rating score) assessment was made. Phase-I was followed by allocation into the groups i.e., study and control groups. In phase-2, a video of surgical procedure was obtained through internet. After all residents have done the procedure initially, 27 participants of the study group were made to watch the videos and learn the steps of procedure while those of the other group did not watch the videos. Participants of both the groups were made to perform the procedure again. GARS (global assessment rating score) was calculated for each individual in their second procedure which included following scores:

1. Respect for tissue
2. Time and motion
3. Instrument Handling
4. Depth perception
5. Bimanual Dexterity All elements scored between 1-5 with a total of 25 score. All procedures were performed under the supervision of a consultant surgeon who was blinded about the groups and make assessment according to the GARS (global assessment rating score).

ELIGIBILITY:
Inclusion Criteria:

* All the postgraduate trainees in surgery and allied specialties
* Age 25 to 35 years
* Both Genders
* Any year of training with at least 3 months of surgical training.

Exclusion Criteria:

* Those residents who did not wish to participate
* Those with less than 3 months of training.
* Consultant surgeons

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
The GARS (global assessment rating score). | 3 Months
  To determine the GARS score of participants before and after watching the procedural video and compare them which include the following
  * Respect for tissue
  * Time and motion
  * Instrument handling
  * Depth perception
  * Bimanual dexterity Total number will be calculated in 2 phases and will be out of 25 and the higher the score, the better the trainee is. The main aspect to be seen will be whether the trainee surgeon improved his GARS score following watching procedural video or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University/PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No